CLINICAL TRIAL: NCT06485908
Title: MEPENDAX: Phase I/II Study of Axitinib (Inlyta®) and Oral Metronomic Etoposide for Pediatric Children and AYA Refractory/Relapsing Medulloblastoma and Ependymoma
Brief Title: Axitinib and Oral Metronomic Etoposide for Pediatric Children and AYA Refractory/Relapsing Medulloblastoma and Ependymoma
Acronym: MEPENDAX
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCAPHM23_0164
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Medulloblastoma; Ependymoma
MeSH Terms: conditions — Medulloblastoma; Ependymoma | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving axitinib in combination with etoposide (Experimental): 1. st stage: Dose escalation The first patient will be included at the level of 1.6 mg/m²/day of axitinib. Patients will be included by cohort of a maximum of 6 patients evaluable for DLT. In the absence of more than 2 patients with DLT during the first 28-day cycle, escalation to the next level will be allowed. Intra-patient dose escalation is not permitted. Non evaluable patients for DLT will be replaced. Six evaluable patients will be enrolled at the last dose level. RP2D will be the DMT or in the absence of DLT the maximum dose evaluated.
     Treatment will be continued until progression, or unacceptable toxicity for a period of 1 year.
     Depending on the number of DLTs observed, a maximum of 18 patients should be included.
  2. nd stage: extension cohort For the second phase of the study, at RP2D, 2 cohorts of 9 patients (ependymoma, medulloblastoma) will be considered in the study. Treatment will be continued until progression, or unacceptable toxicity for a period of 1 year.
  Interventions: Drug: administration of axitinib in combination with etoposide

INTERVENTIONS:
Drug: administration of axitinib in combination with etoposide — 1. st stage:
     * Axitinib (Inlyta®) PO, in the morning and in the evening every day
     * Level -1 : Dose 1.2 mg/m²
     * Level 1: Dose 1.6 mg/m²
     * Level 2: Dose 2.0 mg/m²
     * Level 3: Dose 2.4 mg /m² (equivalent to 4 mg in adults)
     * Etoposide (50 mg capsules or in the form of etoposide phosphate if required): 25 mg/m²/day in the evening orally every day fasting (capped to a maximum of 50 mg/day) First patient will be enrolled at dose level 1
  2. nd stage:
     * Axitinib (Inlyta®) dosing as selected at the 1st stage
     * Etoposide (50 mg capsules or in the form of etoposide phosphate if required): 25 mg/m2/ day in the evening orally every day fasting(capped to a maximum of 50 mg/day)

SUMMARY:
It is an open multicentric phase I/II trial with axitinib (Inlyta®) and metronomic delivery of etoposide for children, adolescent and young adults (AYA) with refractory/ relapsing solid tumors. It is a two-stage trial:

First stage: To determine the Maximum Tolerated Dose (MTD) of the combination of axitinib and oral metronomic etoposide for patient with medulloblastoma or ependymoma Second stage: Extension cohort evaluating the preliminary efficacy at the recommended dose for the phase II (RDP2) of the combination. The 2nd stage will start after a meeting of independent data monitoring committee (IDMC). Two cohorts of 9 patients with ependymoma and medulloblastoma Patients treated at first stage won't be included in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of ependymoma or medulloblastoma
* Methyloma classification performed or available material for methyloma analysis
* Confirmed progressive or refractory disease despite standard therapy, or for which no effective standard therapy exists
* Male and female subjects with > 4 to ≤ 25 years of age at inclusion
* Weight > 20 kg
* Evaluable target lesion(s) according to RAPNO
* Performance status: Karnofsky performance status (for patients >12 years of age) or Lansky Play score (for patients ≤12 years of age) ≥ 70%. Patients who are unable to walk because of paralysis or stable neurological disability, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Life expectancy ≥ 3 months
* No known allergy to any of the compounds in the experimental treatment
* Able to take oral treatments
* Adequate organ function:

Hematologic criteria

* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3 (unsupported)
* Platelet count ≥ 100,000/mm3 (unsupported)
* Hemoglobin ≥ 8.0 g/dL (transfusion is allowed) Cardiac function
* Shortening fraction (SF) >29% and left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography (mandatory only for patients who have received cardiotoxic therapy).

Renal and hepatic function

* Serum creatinine < 1.5 x upper limit of normal (ULN) for age
* Total bilirubin < 1.5 x ULN
* Alanine aminotransferase (ALT)/ Aspartate aminotransferase (AST)/ < 2.5 x ULN

  * Able to comply with scheduled follow-up and with management of toxicity.
  * Females of child bearing potential must have a negative serum pregnancy test within 7 days prior to initiation of treatment.
  * Sexually active patients must agree to use adequate and appropriate contraception (in accordance with Clinical Trials Facilitation and Coordination Group (CTFG) recommendations) while on study drug and for 6 months after stopping the study drug.
  * Patient able to comfortably swallow capsules.
  * Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines.
  * Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.

Non-inclusion Criteria

* Chemotherapy within 21 days of day 1 from the start of study treatment. This period can be shortened in the case of treatment with vincristine (2 weeks) and extended to 6 weeks in the case of treatment with nitrosureas. The period is set to 5 half-lives in the case of targeted therapies or metronomic chemotherapy. The period is set to 2 weeks after bevacizumab administration. Evidence of > Grade 1 recent CNS hemorrhage on the baseline MRI or scan.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
* Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening).
* Known active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
* Presence of any NCI-CTCAE v5 grade ≥ 2 treatment-related extra-hematological toxicity with the exception of alopecia, ototoxicity or peripheral neuropathy.
* Known congenital immunodeficiency.
* Radiotherapy within the 2 months preceding D1 of the start of study treatment. Palliative RT on a non-target lesion is allowed up to 1 weeks before beginning of treatment.
* Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48 hour interval must be maintained before the first dose of the investigational drug is administered.
* Bleeding disorder.
* Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening).
* Known hypersensitivity to any study drug or component of the formulation.
* Absence of effective contraception in patients of childbearing age (see appendix 3)
* Pregnant or nursing (lactating) females.
* Patients with galactose intolerance, lactase deficiency or glucose or galactose malabsorption syndrome (rare hereditary diseases).
* Severe infections requiring parenteral antibiotic therapy.
* Inability to undergo medical monitoring of the trial for geographic, social or psychological reasons.

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | During the first 28 days (cycle 1)
  During first stage
Progression-free survival (PFS) | 3 years (from start of treatment to last follow-up visit)
  During second stage, progression-free survival (PFS) computed as the time interval from the beginning of treatment to the date of centrally-assessed with RAPNO criteria. A central review of all imaging is planned at the end of phase 1 and at the end of phase expansion to evaluate tumor response and progressions. PFS-duration of patients alive free of progression at last follow-up will be censored at the date of last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ANDRE, Principal Investigator — Assistance Publique - Hôpitaux de Marseille